CLINICAL TRIAL: NCT00235222
Title: Evaluation of Viral Efficacy and Safety of a Reduced Dose of Stavudine (d4T): THE PHOENIX STUDY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREPATS 05-01-PHOENIX
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-10

CONDITIONS: HIV
Keywords: Stavudine; Reduced dose of stavudine; Viral load; Peripheral neuropathy; Treatment Experienced
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Stavudine

INTERVENTIONS:
Drug: stavudine

SUMMARY:
Lipodystrophie, peripheral neuropathy and mitochondrial toxicity has been associated to stavudine at standard doses The aim of this study is to evaluate the efficacy of reduced doses of stavudine (30 mg b.i.d.) in HIV patients with controlled viral load and body weight > 60 kg, receiving an antiretroviral therapy containing stavudine 40 mg b.i.d.

DETAILED DESCRIPTION:
Stavudine is a nucleoside inhibitor larged used in HIV treatments and has been associated to mithocondrial toxicity. As it is still largely used in developping countries,the evaluation of reducing dose is of importance.

A single-arm open pilot 48 weeks study to evaluate the capacity of a switch from d4T 40 mg to 30 mg bid in patients with body weight > 60kg to maintain full viral load suppression. Clinical and biological evaluations were carried out at baseline, W24 and W48. Primary end-point is viral load suppression (<400 coies/ml) at W24.

Secondary end-points are : Evolution of CD4 count at W24 and W48, neurological examination at Baseline, W24 and W48, metabolic parameters and stavudine PK at W24.

ELIGIBILITY:
Inclusion Criteria:

* HIV patients
* Patients with an antiretroviral treatment containing stavudine at standard doses (40mg BID) for at least 3 months
* Patients with viral load < 400 copies/ml for at least 3 months

Exclusion Criteria:

* Patients receiving an antiretroviral therapy containing stavudine at 30mg BID
* Current Opportunistic Infection
* Current chemotherapy or under cytokines treatment (PEG, INF, IL2)
* Pregnant or feeding Women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57
Dates: Start 2004-06; Study Completion 2006-03

PRIMARY OUTCOMES:
Proportion of patients with viral load < 400 copies/ml at week S24

SECONDARY OUTCOMES:
Clinical and biological safety of the reduced doses of stavudine at week 24. Percentage of patients with viral load < 400 copies/ml at week 48, evolution of Cd4 count from baseline to W24 and 48. Evolution of metabolic parameters from baseline to W24 and

CONTACTS AND LOCATIONS:
Overall Officials: Manuela BONMARCHAND, MD, Study Chair — Service de médecine Interne Hôpital Pitié Salpêtrière; Hocine AIT-MOHAND, MD, Study Chair — Service de Maladies Infectieuses Hôpital Pitié Salpêtrière
Locations (1):
- Service de Maladies Infectieuses Hôpital Pitié-Salpêtrière, Paris, France